CLINICAL TRIAL: NCT07207811
Title: CLEOPATTRA: Effects of NNC6019-0001 Versus Placebo on Cardiovascular Outcomes in Participants With Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Brief Title: CLEOPATTRA: A Research Study to Look at the Effects of Treatment With a Medicine Called Coramitug (NNC6019-0001) in People With Heart Failure Due to Transthyretin Amyloid (ATTR) Amyloidosis
Acronym: CLEOPATTRA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6019-4958; U1111-1315-5366 (Other: World Health Organization (WHO)); 2024-518899-31 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-09-23; First posted 2025-10-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Amyloid Cardiomyopathy (ATTR CM)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC6019-0001 (Experimental): Participants will receive NNC6019-0001 intravenously (IV). Participants will also have the option to continue any Standard of care (SoC) treatments as recommended by their medical health professional.
  Interventions: Drug: NNC6019-0001
- Placebo (Placebo Comparator): Participants will receive placebo matched to NNC6019-0001 IV. Participants will also have the option to continue any SoC treatments as recommended by their medical health professional.
  Interventions: Drug: Placebo (NNC6019-0001)

INTERVENTIONS:
Drug: NNC6019-0001 — NNC6019-0001 will be administered IV.
  Arms: NNC6019-0001
Drug: Placebo (NNC6019-0001) — Placebo matched to NNC6019-0001 will be administered IV.
  Arms: Placebo

SUMMARY:
This study will find out if a new medicine called NNC6019-0001 can help reduce the risk of heart-related death and illness in participants with a condition called transthyretin amyloid cardiomyopathy (ATTR-CM), which affects the heart. Participants will either receive NNC6019-0001 or a placebo (a treatment with no active medicine), and which one they get is decided by chance. Everyone in the study will continue receiving their usual heart treatments as recommended by their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 18 years or above at the time of signing the informed consent.
* Have an established diagnosis of ATTR-CM (wild-type ATTR [ATTRwt] or variant ATTR [ATTRv]), with cardiac amyloid infiltration, increased left ventricular (LV) wall thickness, and HF.

Note: Target ATTRv recruitment is approximately 15 percent of the study population.

1. Cardiac amyloid infiltration demonstrated by:

   * Cardiac biopsy positive for TTR amyloid, OR
   * Grade 2 or 3 cardiac uptake at pyrophosphate (PYP)/diphosphono-1,2-propanodicarboxylic acid (DPD)/ hydroxymethylene diphosphonate (HMDP) scintigraphy with single-photon emission computed tomography (SPECT/CT) combined with an extracardiac biopsy positive for TTR amyloid, OR
   * Grade 2 or 3 cardiac uptake at PYP/DPD/HMDP scintigraphy with SPECT/CT combined with normal serum free light chain ratio, and negative serum and urine protein electrophoresis with immunofixation (SPIE & UPIE).

   Notes:
   * Non-invasive diagnostic pathway will be confirmed by a centralised expert review.
   * Bone tracer scintigraphy will be conducted using 99m-technetium (Tc)-labelled pyrophosphate (99mTc-PYP), 99mTc-labelled 3,3-diphosphono-1,2-propanodicarboxylic acid (99mTc-DPD), or 99mTc-labeled hydroxymethylene diphosphonate (99mTc-HMDP).
2. Increased LV wall thickness, as assessed by centralised review of echocardiography, showing interventricular septal wall thickness greater than or equal to 12 millimeter (mm).
3. Chronic HF (New York Heart Association [NYHA] Class I-IV) requiring ongoing treatment with a loop diuretic with:

   * At least 1 documented hospitalisation for HF, OR
   * History of HF manifested by signs or symptoms of volume overload or elevated intracardiac pressures (e.g., elevated jugular venous pressure, shortness of breath, signs of pulmonary congestion on x-ray or auscultation, or peripheral oedema).
   * Expected to be on stable cardiovascular medical therapy (defined as no greater than 50 percent dose adjustment and no categorical changes of medications), with the exception of diuretics, 4 weeks prior to the randomisation visit.
   * Completed more than 50 meters on the 6MWT at screening.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Current or previous participation (dosing with active treatment) in a study for an investigational ATTR depleting drug or ATTR gene editing therapy.
* Total bilirubin greater than 3 times the upper limit of normal (ULN) at screening.
* Current diagnosis or history of amyloid light chain, other non-ATTR amyloidosis, known leptomeningeal amyloidosis, or multiple myeloma.
* HF not primarily caused by ATTR-CM (e.g., due to hypertension, valvular heart disease, or ischemic heart disease in the opinion of the investigator).
* Currently hospitalised or hospitalised within 14 days prior to screening.
* Currently treated with positive inotropic medication.
* Uncorrected, severe, haemodynamically significant, left-sided heart valve disease.

Note: Pre-existing echocardiogram up to 2 years old may be used.

* Acute coronary syndrome, unstable angina, stroke, transient ischemic attack, coronary revascularisation, cardiac device implantation, cardiac valve repair, or major surgery within 60 days of screening.
* Prior solid organ transplant or planned solid organ transplant during the study.
* Left ventricular ejection fraction (LVEF) less than 30 percent as assessed by centralised review of echocardiography.
* Presence or history of malignant neoplasm (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, carcinoma in situ/high-grade prostatic intraepithelial neoplasia [PIN], low-risk prostate cancer, or on stable therapy for prostate cancer) within 3 years before screening.
* End-stage renal disease (estimated glomerular filtration rate [eGFR] less than 15 mL/min/1.73 m^2 at screening, or chronic/intermittent haemodialysis or peritoneal dialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2029-06-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences of composite endpoint of cardiovascular (CV) deaths and recurrent CV events (CV hospitalisations and urgent heart failure [HF] visits) | From baseline (week 0) to end of study (EOS) (up to approximately 4 years)
  Measured as count of events.

SECONDARY OUTCOMES:
Change in Kansas city cardiomyopathy questionnaire- clinical summary score (KCCQ-CSS) | From baseline (week 0) to approximately 2 years
  Measured as score on a scale. KCCQ-CSS is a score derived from a 23-item patient-reported outcome (PRO) measure assessing health status in individuals with HF. The score ranges from 0 to 100, with higher scores indicating better health status.
Change in Kansas city cardiomyopathy questionnaire- overall summary score (KCCQ-OSS) | From baseline (week 0) to approximately 2 years
  Measured as score on a scale. KCCQ-OSS is a score derived from a 23-item PRO measure assessing health status in individuals with HF. The score ranges from 0 to 100, with higher scores indicating better health status.
Change in 6-minute walk distance (6MWD) | From baseline (week 0) to approximately 2 years
  Measured in meters.
Number of occurrences of CV events (CV hospitalisation and urgent HF visits) | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured as count of events.
Time to occurrence of CV death | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured in months.
Time to occurrence of all-cause death | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured in months.
Time to first occurrence of composite CKD endpoint: CV death, onset of a persistent decline in eGFR of ≥30% from baseline, onset of a persistent eGFR <15 mL/min/1.73 m^2, or initiation of chronic KRT, including dialysis or kidney transplantation | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured in months. Composite chronic kidney disease (CKD) endpoint comprised of (1) CV death, (2) onset of a persistent decline in estimated glomerular filtration rate (eGFR) of greater than or equal to 30 percent (%) from baseline, (3) onset of a persistent eGFR less than or equal to 15 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2), or (4) initiation of chronic kidney replacement therapy (KRT), including dialysis or kidney transplantation.
Time to hospitalisation due to HF or urgent HF visit | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured in months.
Time to CV events (CV hospitalisation and urgent HF visit) | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured in months.
Number of occurrences of composite endpoint of CV deaths and recurrent CV events (CV hospitalisation, urgent HF visits, and outpatient HF visits) | From baseline (week 0) to EOS (up to approximately 4 years)
  Measured as count of events.
Participant achieving threshold for clinically meaningful within-patient change from the participant's perspective in KCCQ-CSS | From baseline (week 0) to approximately 2 years
  Measured as count of participants.
Participant achieving threshold for clinically meaningful within-patient change from the participant's perspective in KCCQ-OSS | From baseline (week 0) to approximately 2 years
  Measured as count of participants.
Participant achieving threshold for clinically meaningful within-patient change from the participant's perspective in 6-minute walk test (6MWT) | From baseline (week 0) to approximately 2 years
  Measured as count of participants.
Change in stroke volume (SV) | From baseline (week 0) to week 52
  Measured in milliliter (mL).
Change in N-terminal pro B-type natriuretic peptide (NT-proBNP) | From baseline (week 0) to week 52
  Measured as ratio to baseline.
Change in high-sensitivity (hs) troponin I | From baseline (week 0) to week 52
  Measured in nanograms per milliliter (ng/mL).
Change in troponin T | From baseline (week 0) to week 52
  Measured in ng/mL.
Hierarchical composite of time to all-cause death as assessed by the win ratio | From baseline (week 0) up to approximately 2 years
  Measured as total wins for each treatment group.
Hierarchical composite of number of CV events (CV hospitalisations or urgent HF visits) as assessed by the win ratio | From baseline (week 0) up to approximately 2 years
  Measured as total wins for each treatment group.
Hierarchical composite of difference > 15, > 10 and > 5 points in KCCQ-OSS as assessed by the win ratio | From baseline (Week 0) to approximately 2 years
  Measured as total wins for each treatment group.
Hierarchical composite of difference > 70 and > 30 meters in 6-minute walk test (6MWT) as assessed by the win ratio | From baseline (Week 0) to approximately 2 years
  Measured as total wins for each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (276):
- United States (62):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of California San Diego (UCSD) - Sulpizio Cardiovascular Center (SCVC), La Jolla, California
  - Keck School of Medicine USC - Healthcare Consultation Center 2 (HCCII), Los Angeles, California
  - UCI Medical Center, Orange, California
  - Profound Research LLC at Southern California Heart Specialists, Pasadena, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Northbay Cardiology Inc., Santa Rosa, California
  - Lucile Packard Children's Hospital, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Heart & Vascular Institute (MHVI) - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Heart and Vascular Hospital, Gainesville, Florida
  - Northeast Georgia Heart Center, Pc (Nghc), Gainesville, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University Clinical and Translational Sciences Institute, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - Endeavor Health - Glenbrook Hospital, Glenview, Illinois
  - Indiana University (IU) Health - Methodist Professional Center II, Indianapolis, Indiana
  - LCMC - LSU University Medical Center New Orleans LCMC Center, New Orleans, Louisiana
  - University of Maryland Medical Center (UMMC) - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Maryland Medical Center (UMMC), Baltimore, Maryland
  - John Hopkins Medicine, Baltimore, Maryland
  - Tufts Medical Center (TMC) - Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Profound Research, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cardiology Associates Research, LLc, Tupelo, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore University Hospital, Northwell Health, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Laurelton Heart Specialist, PC, Rosedale, New York
  - Yeshiva University - Albert Einstein College of Medicine - Montefiore Medical Center (MMC), The Bronx, New York
  - Duke University Health System, Durham, North Carolina
  - The Carl and Edyth Lindner-Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Abington Hospital - Jefferson Health, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Milton S.Hershey Medical Center - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) - Center for Image-Guided Neurosurgery, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Saint Thomas Health, Nashville, Tennessee
  - Ascension Seton Heart Institute - Medical Park Tower Location, Austin, Texas
  - St. Davids Heart and Vascular, Austin, Texas
  - Baylor Scott & White Research Institute - Annette C. and Harold C. Simmons Transplant Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor St. Luke Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott & White The Heart Hospital, Plano, Texas
  - Inova Fairfax Hospital - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
- Australia (13):
  - ST Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Liverpool Renal Clinical Research Centre, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Advara HeartCare - Milton, Milton, Queensland
  - Metro South Health - Princess Alexandra Hospital (PAH), Woolloongabba, Queensland
  - Central Adelaide Local Health Network - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Private Hospital, Adelaide, South Australia
  - Advara HeartCare - Leabrook, Leabrook, South Australia
  - Hobart Hospital-Royal Hobart Hospital, Hobart, Tasmania
  - Victorian Heart Hospital, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Joondalup Cardiovascular Trials Foundation Inc., Joondalup, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (11):
  - Hopital Universitaire de Bruxelles/ Academisch Ziekenhuis Brussel, Brussels, Anderlecht
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - Universitair Ziekenhuis Brussel, Jette, Brusselss
  - ZOL Genk, Campus Sint-Jan, Waterschei-Zwartberg, Limburg
  - AZORG Ziekenhuis, Aalst, Oost-Vlaanderen
  - Algemeen Ziekenhuis Sint-Blasius (AZSB), Sint-Gillis-Dendermonde, Oost-Vlaanderen
  - Az Middelheim, Antwerp
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Regional CHR de la Citadelle, Liège
  - Clinique Universitaire de Mont Godinne, Yvoir
- Brazil (16):
  - Instituto D'Or de Pesquisa e Ensino - Hospital Cardio Pulmonar (HCP), Salvador, Estado de Bahia
  - L2 IP - Instituto de Pesquisas Clinicas LTDA, Brasília, Federal District
  - Cardresearch Cardiologia Assistencial e de Pesquisa Ltda, Belo Horizonte, Minas Gerais
  - NUPEC Cardio, Belo Horizonte, Minas Gerais
  - Eurolatino Pesquisas Medicas Ltda - (Eurolatino Medical Research - EMR), Uberlândia, Minas Gerais
  - Pontificia Universidade Catolica do Parana (PUCPR) - Centro de Ciencias Biologicas e da Saude (CCBS), Curitiba, Paraná
  - Instituto D'Or de Pesquisa e Ensino - Recife, Recife - PE, Recife - PE
  - Universidade de Caxias do sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual de Campinas - UNICAMP, Campinas, São Paulo
  - Synvia Laboratórios e Toxicologia Ltda - Synvia Clinical, Campinas, São Paulo
  - Centro Avancado de Pesquisa-Estudo para-Diagnostico-CAPED, Ribeirão Preto, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina De Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Instituto de Cardiologia Dante Pazzanese, São Paulo
  - Pseg Centro De Pesquisa Clinica S.A, São Paulo
  - Universidade de Sao Paulo (USP) Hospital das Clinicas da Faculdade de Medicina (HCFMUSP), São Paulo
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - CIUSSS du Saguenay Lac-Saint-Jean, Québec, Chicoutimi
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Health Sciences North Research Institute-Advanced Medical Research Institute of Canada, Greater Sudbury, Ontario
  - Cardio Health Clinical Trials, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Cardio Health Clinical Trials, Mississauga, Ontario
  - Cardiohealth Medical Clinic, Scarborough Village, Ontario
  - Riverside Cardiology and Diagnostic Imaging, Toronto, Ontario
  - Hotel Dieu de Quebec, Québec
- China (31):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - FuWai Hospital, CAMS & PUMC, Beijing, Beijing Municipality
  - Beijing University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - China-Japan Union Hospital, Changchun, Changchun
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Southern Medical University, Guangzhou, Guangdong
  - Guangdong Academy of Medical Science (GAMS) - Guangdong General Hospital (GGH) - Guangdong Neuroscience Institute, Guangzhou, Guangdong
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huazhong University of Science and Technology - Tongji Medical College - Tongji Hospital, Wuhan, Hubei
  - Wuhan University - Renmin Hospital (Hubei General Hospital), Wuhan, Hubei
  - Xiangya Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Medical University (NMU) - Jiangsu Province Hospital (First Affiliated Hospital), Nanjing, Jiangsu
  - Shengjing University Of China Medical University, Liaoning, Liaoning
  - Qi-Lu Hospital of Shandong University School of Medicine, Jinan, Shandong
  - Shandong University School of Medicine - Shandong Provincial Hospital (SPH), Jinan, Shandong
  - Renji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University (SJTU) - Shanghai Chest Hospital (SCH), Shanghaishi, Shanghai Municipality
  - Shanxi Medical University - First Hospital, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - TEDA Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, School of Medicine, ZheJiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital Of Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital Of Nanchang University, Nanchang
- Czechia (7):
  - Edumed s.r.o., Broumov, Královéhradecký kraj
  - St. Anne''s University Hospital / International Clinical research Centre, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
  - Interni klinika kardiologie a angiologie 1. Lekarske fakulty a Vseobecne fakultni nemocnice v Praze, Prague
  - IKEM, Kardiologicka klinika, Prague
  - Kardiologie-MUDr. Antonin Dufka, Uherské Hradiště
- Denmark (3):
  - Hjertecentret (The Heart Center)-Copenhagen University Hospital/Rigshosptalet, Copenhagen, Capital Region
  - Aarhus Universitetshospital Skejby, Aarhus, Central Jutland
  - Odense Universitetshospital, Odense C
- France (19):
  - Centre Hospitalier Universitaire d'Amiens-Picardie - Site Sud, Amiens
  - Centre Hospital Regional Et Universitaire De Tours (Chru Tours) - Houpital Trousseau, Chambray-lès-Tours
  - Hospital Henri Mondor, Créteil
  - CHU De Dijon Hopital Du Bocage, Dijon
  - Centre Hospitalier Departemental Vendee (CHD) - L'Hopital de la Roche-sur-Yon (CHD Les Oudairies), La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Grenoble (CHUG) Hopital Nord, La Tronche
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital de La Timone, Marseille
  - Hospital Center Annecy Genevois-Centre Hospitalier de la Region d'Annecy CHRA, Metz-Tessy
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier Arnaud de Villeneuve, Montpellier
  - CHU De Nantes - Hopital Laennec, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Groupement Hospitalier Universitaire Ouest - Hopital Europeen Georges-Pompidou (HEGP), Paris
  - Hopital Bichat - Claude-Bernard, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers la Miletrie, Poitiers
  - Centre Hospitalier Universitaire (CHU) de Rennes, Rennes
  - Centre Hospitalier de Toulon - Hopital Sainte-Musse, Toulon
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital Rangueil, Toulouse
  - Private Hospital Medipole, Villeurbanne
- Germany (13):
  - Universitätsklinik Der Ruhr-Universität Bochum, Bad Oeynhausen
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Klinikum Bielefeld Mitte, Bielefeld
  - Universitaetsklinikum Koeln, Cologne
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - University Heart Center Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - University of Munich (LMU)-Grosshadern Hospital, Munich
  - Deutsches Herzzentrum Muenchen, München
  - Universitaetsklinikum Muenster, Münster
  - University of Wurzburg, Comprehensive Heart Failure Center (CHFC), Würzburg
- Italy (24):
  - Policlinico S.Orsola Malpighi, Universita di Bologna, Bologna
  - Azienda Sanitaria del Sudtirol-Ospedale di Bolzano, Bolzano
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Policlinico Gaspare Rodolico - San Marco, Catania
  - Azienda Ospedaliera Universitaria Di Ferrara, Cona
  - Universita Degli Studi Di Firenze - Azienda Ospedaliero-Universitaria Careggi (AOUC), Florence
  - Ospedale di Ivrea, Ivrea
  - ASST di Lecco - Presidio Ospedaliero A. Manzoni di Lecco, Lecco
  - Azienda Ospedaliera Universitaria Gaetano Martino Messina, Messina
  - Fondazione Irccs Ca' Granda Ospedale Maggioe Policlinico Di Milano, Milan
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan
  - Centro Cardiologico Monzino IRCCS, Milan
  - Azienda Ospedaliera San Paolo - Universita Degli Studi Di Milano, Milan
  - Istituto Auxologico Italiano, IRCCS, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera dei Colli - Ospedale Monaldi, Napoli
  - Divisione di Cardiologia con Utic ed Emodinamica, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Amyloidosis Research & Treatment Center, Fondazione Irccs Policlinico San Matteo, Pavia
  - Universita degli Studi di Perugia, Perugia
  - Fondazione Toscana Gabriele Monasterio Per La Ricerca Medica E Di Sanita Pubblica (Ftgm), Pisa
  - Istituto Patologia Speciale Medica Universita Cattolica del Sacro Cuore - Policlinico Universitario Agostino Gemelli, Rome
  - Ospedale Sant'Andrea Hospital, Rome
  - Polo Cardiologico - Ospedale Cattinara (ASUGI), Trieste
- Japan (25):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Instituto D'Or de Pesquisa e Ensino - Hospital Cardio Pulmonar (HCP), Salvador, Brazil
  - Uwajima City Hospital, Uwajima-shi, Ehime
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Hospital of University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Kurume University - Research Center for Innovative Cancer Therapy, Kurume-shi, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaid
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Mie University Hospital, Tsu, Mie-ken
  - Shinshu University Hospital, Shinshu University Graduate School Of Medicine, Matsumoto, Nagano
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Nara Medical University Hospital, Kashihara, Nara
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Yamaguchi University Hospital, Yamaguchi Prefecture, Yamaguchi
  - Kitasato University - Kitasato University Hospital (KUH), Kanagawa
  - Social Welfare Organization Imperial Gift Foundation, Inc. Saiseikai Kumamoto Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Keio University Hospital, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
- Netherlands (4):
  - Erasmus Medisch Centrum 1, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center (MUMC), Maastricht
  - Universitair Medisch Centrum Utrecht (UMC Utrecht), Utrecht
- South Korea (7):
  - Seoul National University Bundang Hospital (SNUBH), Seongnam-si, Gyeonggi-do
  - Inje University Haeundae Paik Hospital, Busan
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (21):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitari Germans Trias i Pujol (HUGTP), Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Son Llatzer (HSLL), Palma de Mallorca
  - Hospital Clinico Universitario De Santiago De Compostela, Santiago de Compostela
  - Universidad de Sevilla - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Servicio Andaluz de Salud (SAS) - Hospital San Juan de la Cruz, Úbeda
  - Fundacion Investigacion Clinico de Valencia (FIHCUV) - Instituto de Investigacion Sanitaria (INCLIVA), Valencia
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
  - Hospital Clinico Universitario Lozano Blesa de Zaragoza, Zaragoza
- United Kingdom (9):
  - The Royal Free Hospital - Royal Free London NHS Foundation Trust, London, Greater London
  - Synexus Manchester Clinical Research Centre, Manchester, Greater Manchester
  - Synexus Scotland Clinical Research Centre, Bellshill, Lanarkshire
  - Synexus North East Clinical Research Centre, Hexham, Northumberland
  - Synexus Midlands Clinical Research Centre, Birmingham, West Midlands
  - Velocity Clinical Research, Bristol, Bristol
  - Synexus Wales Clinical Research Centre, Cardiff
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Richmond Pharmacology - MHRA Phase 1 Unit, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com